CLINICAL TRIAL: NCT05307367
Title: Identifying Molecular Factors Contributing to Cancer-associated Muscle Mass Loss and Providing Clinical Evidence for Exercise Mechanisms to Functionally Restore Muscle in Cancer
Brief Title: Cancer-associated Muscle Mass - Molecular Factors and Exercise Mechanisms
Acronym: PANACEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2447473
Record Dates: First submitted 2022-01-25; First posted 2022-04-01 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-01

CONDITIONS: Cachexia; Neoplasms; Exercise; Metabolism; Body Composition; Insulin Resistance; Physical Functional Performance; Quality of Life; Sarcopenia; Caregivers; Adipose Tissue; Muscle, Skeletal; Patient Reported Outcome Measures; Gastrointestinal Microbiome; Proteomics; Lipidomics; Epigenomics; Mitochondria
MeSH Terms: conditions — Cachexia; Neoplasms; Motor Activity; Insulin Resistance; Sarcopenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: WP1+2: longitudinal research design of 80 patients with newly diagnosed non-small cell lung cancer, over 12 weeks registration of biomedical variables incl. blood samples, physical performance, body composition, and patient- and caregiver-reported outcomes. On a subgroup in WP2 (n=40) obtaining skeletal muscle biopises, adipose tissue (AT) biopsies, and peripheral blood samples before and after 12 weeks of 1st line treatment. In WP2 40 healthy matched controls will be assessed as well.
  WP3: a interventional study where 24 patients in active treatment for NSCLC will participate in a 8 weeks one-leg exercise training. The design has an important advantage that the contralateral leg is an untrained control. In WP3 24 healthy matched controls will be assessed as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WP1-3 (Experimental): WP1+2: no intervention WP3: exercise training as intervention
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Patients will be enrolled in a 8 week, supervised, single-leg kicking training intervention (1h, or as long as possible, 60-70% peak workload (PWL), 2-5 days a week). Healthy age-, body weight-, gender- and activity level-matched control subjects will undertake the intervention matched to the %PWL obtained by the patients who complete the study.

SUMMARY:
Muscle mass loss is a common adverse effect of cancer. Muscle mass loss occurs with or without reduction in body weight. Cancer cachexia (CC) is the involuntary loss of body weight of >5% within 6 months and it occurs in 50-80% of patients with metastatic cancer.

It is estimated that CC is a direct cause of up to 30% of all cancer-related deaths. No treatment currently is available to prevent CC, likely because the chemical reactions that causes of this devastating phenomenon in unknown.

No treatment currently is available to prevent muscle mass loss in patients with cancer but is urgently needed as the reduced muscle mass and function is associated with impaired physical function, reduced tolerance to anticancer therapy, poor quality of life (QoL), and reduced survival. There is evidence of an interdependence between informal caregiver (e.g. spouse) and patient QoL. Thus, identifying caregiver distress and needs can potentially benefit QoL for patients with cancer cachexia. Despite the enormous impact on disease outcomes, it is not known why the loss of muscle mass and function occurs and very few studies have investigated the underlying molecular causes in humans. In particular, there is a severe lack of studies that have obtained human skeletal muscle and adipose tissue sample material. Such reference sample materials will be invaluable to obtaining in-depth molecular information about the underlying molecular causes of the involuntary but common muscle mass and fat mass loss in cancer.

At a whole body level, cancer cachexia is associated with reduced sensitivity to the hormone insulin, high levels of lipids in the blood, and inflammation. Within the skeletal muscle, the muscle mass loss is associated with elevated protein breakdown and reduced protein build-up while emerging, yet, limited data also suggest malfunction of the power plants of the cells called mitochondrions. The role of malnutrition and how it contributes to weight loss is understood only to the extent of the observed loss of appetite and the reduced food intake because of pain, nausea, candidiasis of the mouth, and breathlessness. Evidence is increasing that the environment of the intestinal system could be implicated in cancer cachexia, yet, the possible effect of cancer and the cancer treatment on the intestinal environment is not understood. Thus, large and as yet poorly understood details of this syndrome precede a later weight loss.

Exercise training could help restore muscle function and how the chemical reactions works in cancer. In healthy people, and patients with diabetes, cardiovascular disease, and obesity exercise potently improves health. Exercise has been thought to slow down the unwanted effects of cancer cachexia by changing the reactions mentioned above. Thus, there is a tremendous gap in our knowledge of how and if exercise can restore the cells power plants function, muscle mass, strength, and hormone sensitivity in human cachexic skeletal muscle. Tackling that problem and examining potential mechanisms, will enable us to harness the benefits of exercise for optimizing the treatment of patients with cancer.

The data will provide novel clinical knowledge on cachexia in cancer and therefore addressing a fundamental societal problem.

Three specific aims will be addressed in corresponding work packages (WPs):

* investigate the involvement of hormone sensitivity of insulin and measure the chemical reactions between the cells in patients with lung cancer (NSCLC) and describe the physical performance and measure amount of e.g. muscles and adipose tissue across the 1st type of cancer treatment and understand how that is related to the disease and how patients and informal caregiver feel (WP1).
* find changes in the chemical reactions in skeletal muscle, adipose tissue (AT), and blood samples in these patients, to understand how to predict how the disease will develop (WP2).
* measure changes of skeletal muscle tissue in response to exercise and see if it might reverse the hormone insensitivity and improve muscle signaling and function (WP3).

The investigators believe that:

* the majority of patients with advanced lung cancer, at the time of diagnosis already are in a cachectic state, where they lose appetite, and have hormonal changes, and an overall altered chemical actions between the cells affecting both muscle mass and AT. The investigators propose that all this can predict how the disease will progress, and how patient- and informal caregiver fell and how they rate their quality of life.
* lung cancer and the treatment thereof is linked with changes in the blood, the muscle tissues, and the adipose tissues, especially in patients experiencing cachexia, that could be targeted to develop new treatment.
* exercise can restore the muscles and improve insulin sensitivity and improve the function of the cells power plants in patients with lung cancer-associated muscle problems.

ELIGIBILITY:
Inclusion Criteria, WP1+WP2X+WP2:

* Men and women at or above the age of 18
* Histological and radiological verified NSCLC (both squamous and adenocarcinoma) st. IIIb/IV stage not eligible to concurrent chemo/radiation therapy as primary treatment
* Referred for 1st line palliative anticancer therapy (platin based, immunotherapy, combined therapy or TKI), this goes for WP1 + WP2
* Referred for palliative anticancer therapy (platin based, immunotherapy, combined therapy or TKI), for recurrent cancer, this goes only for WP2X.
* Having a staging/baseline CT within 4 weeks of initiation of treatment (PET/CT are also allowed), or a baseline scan planned within the first week of treatment.
* ECOG Performance Status 0-2
* Having signed the informed consent form

Exclusion Criteria, WP1+WP2X+WP2:

* Any other known malignancy requiring active treatment (prior cancer diagnosis is not some exclusion criteria if oncology-treatment is completed)
* Local palliative radiotherapy as primary treatment
* ECOG Performance status > 2
* Physical disabilities excluding physical testing
* Inability to understand Danish
* Inability to understand scoring systems/patient-reported outcome measures

Inclusion Criteria, WP3:

* Men and women above the age of 18
* Histological and radiological verified NSCLC (both squamous and adenocarcinoma) st. IIIb/IV stage
* ECOG Performance Status 0-2
* Having signed the informed consent form.

Exclusion Criteria, WP3:

* Any other known malignancy requiring active treatment (prior cancer diagnosis is not some exclusion criteria if oncology-treatment is completed)
* ECOG Performance Status > 2
* Physical disabilities excluding physical testing
* Inability to understand Danish
* Inability to understand scoring systems/patient-reported outcome measures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Disease outcome | 12 weeks
  according to RECIST criteria where disease status is placed into four different groups (Complete Response, Partial Response, Stable Disease, or Progressive Disease)
Muscle mass | 12 weeks
  changes in L3 CT-derived skeletal muscle index (SMI) (cm2/m2)

SECONDARY OUTCOMES:
Insulin sensitivity status | 8 weeks
  Glucose infusion rate during the hyperinsulinemic euglycemic clamp to ascertai the insulin sensitivity
Proteomic changes in skeletal muscle | 12 weeks
  Skeletal muscle biopsies from vastus lateralis muscle will be analyzed using mass spectronomy to determine proteomic chances in response to non-small cell lung cancer in skeletal muscle.
Patient-reported Quality-of-Life (QoL) | 12 weeks
  Total Quality-of-Life score on The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30. Fom 1 (very poor) to 7 (excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Lykke Sylow, Ass.proff., Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, DK, Denmark